CLINICAL TRIAL: NCT03570866
Title: Positron Emission Tomography and Computed Tomography in the Management of Early Stage Intermediate and High-risk Endometrial Cancer
Brief Title: PET/CT in the Management of Patients With Early Stage Endometrial Cancer
Acronym: ENCA-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: ENCA-1
Record Dates: First submitted 2018-05-31; First posted 2018-06-27 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Endometrium Cancer
Keywords: Endometrial cancer; Positron emission tomography
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Positron Emission Tomography Computed Tomography; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early stage endometrial cancer: Women with diagnosis of intermediate and high-risk early stage endometrial cancer.
  Interventions: Diagnostic Test: Positron emission tomography and computed tomography; Procedure: Surgical treatment

INTERVENTIONS:
Diagnostic Test: Positron emission tomography and computed tomography — Preoperative staging of early stage intermediate and high-risk endometrial cancer with positron emission tomography and computed tomography.
Procedure: Surgical treatment — Surgical treatment of early stage intermediate and high-risk endometrial cancer by usual practice: peritoneal cytology, total abdominal hysterectomy, bilateral salpingo-oophorectomy, systematic pelvic and para-aortic lymphadenectomy.

SUMMARY:
Endometrial cancer (EC) is the most common gynecologic malignancy in the developed countries and is the fifth most common cancer among women worldwide. Typically present well or moderately differentiated, early stage endometrioid histotype with a prognosis usually favorable. Pelvic lymph nodes (LNs) represent the most common site of extra-uterine disease in patients with clinical early stage disease and the role of lymphadenectomy in early stage EC has been one of the major controversies in gynecology oncology. Lymphadenectomy doesn't improve survival or reduce disease recurrence although supported to provide prognostic information and allowing tailoring of adjuvant therapy. Nevertheless, lymphadenectomy is not performed without serious short-term and long-term morbidity. Although surgical staging is the most accurate and standard method to determine LNs involvement, the introduction in clinical practice of a non-invasive modality that allows an accurate staging of EC would be essential. Available evidence report the accuracy of Positron Emission Tomography and Computed Tomography (PET/CT) for the detection of LN metastasis in EC with a sensitivity of 63% and specificity of 94.7%. This prospective comparative analysis between PET/CT, histological findings, and follow up data will be performed to investigate the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of integrated PET/CT for nodal staging of EC per patient and per LN chain analyses, in women affected by intermediate (grade 1 and 2 endometrioid lesions with deep myometrial invasion > 50% or grade 3 endometrioid lesion with < 50% myometrial invasion) or high risk (grade 3 endometrioid lesion with deep myometrial invasion > 50% or non-endometrioid histotype) early-stage EC. Furthermore, the preoperative classification of EC in intermediate and high-risk class will allow to investigate its prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of early stage intermediate and high-risk endometrial cancer.

Exclusion Criteria:

* Not eligible for standard surgical treatment; Not eligible for preoperative staging with PET/CT

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Woman referred for diagnosis of early stage intermediate and high-risk endometrial cancer that undergo PET/CT staging and standard surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of positron emission tomography and computed tomography | Through study completion, an average of 5 year
  Comparing Positron emission tomography and computed tomography results with Histopathological findings served as the standard of reference. True positive, True negative, False positive, False negative. Sensitivity, Specificity, Negative predictive value, Positive predictive value.

SECONDARY OUTCOMES:
Progression free survival | Through study completion, an average of 5 year
  Events of disease recurrence in the study group
Overall survival | Through study completion, an average of 5 year
  Events of death in the study group

CONTACTS AND LOCATIONS:
Overall Officials: Simone Garzon, M.D., Principal Investigator — Universita di Verona; Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Massimo Franchi, M.D., Principal Investigator — Universita di Verona

IPD SHARING:
Plan to Share IPD: Undecided